CLINICAL TRIAL: NCT04687085
Title: Effects of a Brief Mindful Meditation Intervention on Patient Anxiety and Satisfaction for Labor Epidural Catheter Placement: a Randomized Controlled Trial
Brief Title: Mindful Meditation for Epidural Catheter Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Dominique Arce, Instructor in Anesthesia, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019P003456
Record Dates: First submitted 2020-12-21; First posted 2020-12-29 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neutral Content (Placebo Comparator): Participants will listen to a 10 minute neutral content recording just prior to epidural catheter placement.
  Interventions: Other: 10 minute mindful meditation recording
- Mindful Meditation (Experimental): Participants will listen to a 10 minute mindful meditation recording just prior to epidural catheter placement.
  Interventions: Other: 10 minute mindful meditation recording

INTERVENTIONS:
Other: 10 minute mindful meditation recording — 10 minute mindful meditation recording

SUMMARY:
Given the high prevalence of neuraxial analgesia use during labor and the anxiety associated with these procedures, a method to decrease this anxiety could benefit millions of laboring women each year. Mindfulness practice has been used by many groups to decrease anxiety during pregnancy with optimistic results. However, there has been no major study evaluating the role of mindfulness interventions on anxiety associated with neuraxial placement. The purpose of our study is to address this gap in knowledge.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effects of a brief mindful meditation intervention on anxiety and satisfaction regarding epidural catheter placement for laboring parturients.The investigators hypothesize that a brief mindful meditation intervention, consisting of a 10 minute auditory instructional practice, implemented before epidural catheter placement will:

1. Decrease anxiety
2. Increase satisfaction

compared to a neutral 10 minute auditory recording control, in participants undergoing labor epidural catheter placement.

The secondary objective of this study is to evaluate whether anesthesia providers experience a difference in satisfaction with labor epidural catheter placement in participants who listen to a brief mindful meditation intervention prior to epidural catheter placement. The investigators hypothesize that anesthesia providers placing labor epidural catheters in patients who listen to a brief mindful meditation intervention prior to labor epidural catheter placement will:

1. Experience an increase in satisfaction with labor epidural catheter placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for enrollment if they are greater than 18 years of age, admitted for vaginal delivery, anticipating epidural analgesia, and report a numerical pain scale rating of 3 or less at the time of enrollment.

Exclusion Criteria:

* Do not speak English or admitted for cesarean delivery will be excluded from the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy
Enrollment: 100 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Anxiety level after epidural catheter placement | Measure 1 time, 10 minutes after epidural catheter placement
  Level of anxiety on a numerical rating scale
Pain level after epidural catheter placement | Measure 1 time, 10 minutes after epidural catheter placement
  Level of pain on a numerical rating scale

SECONDARY OUTCOMES:
Provider satisfaction level after epidural catheter placement | Measure 1 time, 10 minutes after epidural catheter placement
  Anesthesia provider placing the epidural catheter satisfaction with placement conditions on a numerical rating scale

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
To maintain privacy and confidentiality, patient data will be labeled with an alphanumeric code, the key to the code will be kept in a secure location separate from other data forms and will only be accessible to the investigators.

REFERENCES:
- [Derived] Lumbreras-Marquez MI, Lazaridou A, Villela-Franyutti D, Fields KG, Farber MK, Nelson ER, Schreiber KL, Arce DY. Mindful meditation for epidural catheter placement during labor: a single-center randomized controlled trial. Pain Med. 2026 Jan 1;27(1):26-32. doi: 10.1093/pm/pnaf075. PMID 40570097